CLINICAL TRIAL: NCT04564456
Title: A Pivotal, Randomized, Single-dose, Open Label, Two-treatment, Two-sequence, Two-period, Crossover Study Under Fasting Conditions to Examine the Bioequivalence Between Fluticasone Propionate 500 mcg and Salmeterol Xinafoate 50 mcg Inhalation Powder/Respirent Pharmaceuticals vs. ADVAIR DISKUS® 500/50 Inhalation Powder/GSK in Healthy Volunteers
Brief Title: A Pivotal Bioequivalence Study Between Fluticasone Propionate 500 mcg and Salmeterol Xinafoate 50 mcg Inhalation Powder/Respirent Pharmaceuticals vs. ADVAIR DISKUS® 500/50 Inhalation Powder/GSK in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respirent Pharmaceuticals Co Ltd. (Industry)
Collaborators: Becro Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BREATH-BE500-PIVOTAL
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Bioequivalence
Keywords: bioequivalence; fluticasone propionate; salmeterol xinafoate; ADVAIR
MeSH Terms: interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Intervention Model Description: One-center crossover, randomized, 2-period, 2-sequence (RT and TR), single dose, laboratory-blinded study
Who Masked: Outcomes Assessor
Masking Description: laboratory-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test Product (Experimental): Fluticasone propionate 500 mcg and salmeterol xinafoate 50 mcg/Respirent Pharmaceuticals
  Interventions: Drug: Fluticasone propionate 500 mcg and salmeterol xinafoate 50 mcg/Respirent
- Reference Product (Active Comparator): ADVAIR DISKUS® 500/50
  Interventions: Drug: ADVAIR DISKUS® 500/50

INTERVENTIONS:
Drug: Fluticasone propionate 500 mcg and salmeterol xinafoate 50 mcg/Respirent — 2 inhalations of Test oproduct in one study period
  Arms: Test Product
Drug: ADVAIR DISKUS® 500/50 — 2 inhalations Reference product in one study period
  Arms: Reference Product

SUMMARY:
Bioequivalence study between two inhaler products of fixed dose combination of fluticasone propionate and salmeterol xinafoate inhalation powder

DETAILED DESCRIPTION:
A bioequivalence study of a single dose of the fixed-dose combination of fluticasone propionate and salmeterol xinafoate inhalation powder administered from Fluticasone propionate 500 mcg and Salmeterol xinafoate 50 mcg inhalation powder/Respirent Pharmaceuticals (test-Τ) as 2 inhalations and ADVAIR DISKUS® 500/50 mcg inhalation powder/GSK (reference-R) in healthy volunteers under fasting conditions. The study will be one-center crossover, randomized, 2-period, 2-sequence (RT and TR), single dose, laboratory-blinded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both genders, aged ≥18 and ≤60 years.
* Subjects with Body Mass Index (ΒΜΙ) ≥18.5 and <30.0 kg/m2.
* Healthy volunteers are declared healthy based on medical history, physical examination, ECG, pulmonary function test (a forced expiratory volume in 1 second (FEV1) ≥80% of the predicted normal value), and clinical laboratory values within the laboratory stated normal range; if not within this range, they must be without any clinical significance according to the Investigator.
* Females who participate in the study are either at reproductive age i.e.pre-menopausal or unable to gestate [i.e. post-menopausal (absence of menses for 12 months prior to drug administration), hysterectomy, bilateral oophorectomy, tubal ligation at least 6 months prior to drug administration].
* Subjects that are non-smokers.
* Subjects that, in the opinion of the principal investigator/medical officer, are able to communicate and comply with the study procedures and protocol restrictions as evidenced by the Informed Consent Form (ICF) duly read, signed and dated by the subject prior to study initiation.
* Subjects able to use the inhalers according to given instructions, as judged by the Investigator or study nurse.

Exclusion Criteria:

* Hypersensitivity to the active substance(s) or to the excipient (lactose which contains small amounts of milk protein may cause allergic reactions) or related class (any sympathomimetic drug or any inhaled, intranasal, or systemic corticosteroid therapy) of the medicinal product
* Clinically significant illness or surgery within four weeks prior to dosing.
* Clinically significant ECG abnormalities or vital sign abnormalities (seated systolic blood pressure <90 or >140 mmHg, seated diastolic blood pressure <50 or >90 mmHg or heart rate less than 50 or over 100 bpm) at screening.
* Clinically significant history or presence of chronic bronchitis, emphysema,asthma or any other lung disease.
* History or presence of pulmonary tuberculosis.
* Viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks prior to the screening visit.
* History or presence of significant cardiovascular, endocrinal, neurologic, immunological, psychiatric or metabolic disease.
* History of significant alcohol or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to screening visit (more than 14 alcohol units per week) [1Unit =150 ml of wine, 360 ml of beer, or 45 ml of 40% alcohol].
* Inability to abstain from alcohol for the duration of study period.
* Presence of disease markers for Hepatitis B, Hepatitis C or HIV at screening.
* Positive results for drugs of abuse (barbiturates, marijuana, opioids, benzodiazepines and methadone) in saliva before each administration.
* Positive alcohol breath test before each administration.
* Use of soft drugs (such as marijuana) within three months prior to screening or hard drugs such as crack, cocaine or heroin within one year prior to screening visit
* Intake of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers are barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors are, erythromycin, ketoconazole, indinavir, cobicistat-containing products) within one month prior to administration of the study medication. Under these circumstances, subject inclusion will be judged by the principal investigator.
* History of peptic ulcer, other gastrointestinal disorders (e.g. chronic diarrhoea, irritable bowel syndrome) or unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting) or significant hepatic, renal or other condition that is known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Use of oral or parenteral corticosteroids in the previous four 4 weeks
* Eye disorders especially Glaucoma (or a family history of glaucoma)
* Use of prescription medication (within 14 days prior to the first administration of study medication) or over-the-counter (OTC) products (including food supplements vitamins and herbal supplements) within one week (7 days) prior to the first administration of study medication, except for topical products without systematic absorption. Contraceptives are allowed.
* Vaccination for prophylaxis from seasonal flu or any other vaccination within seven days prior to administration
* History of allergy to any food, intolerance or special diet, that in the opinion of the medical sub-investigator could contraindicate the subject's participation in the study.
* A depot injection or an implant of any drug (except hormonal contraceptives) within 3 months prior to treatment administration.
* Donation of plasma (500 ml) within 7 days prior to treatment administration.
* Donation of whole blood or loss of whole blood ≥ 500 ml prior to administration of the study medication within 30 days prior to treatment administration.
* Participation in another clinical trial simultaneously.
* Subjects receiving special diet or having intolerance in any of the provided study meals or refusing to eat the study meals
* Application of tattoo or body piercing within 30 days prior to treatment administration.
* Non-tolerance to venipuncture.
* Breastfeeding women.
* Positive pregnancy test at screening
* Females of reproductive age that had sexual intercourse with a non-sterile male partner without protection within 14 days prior to drug administration

Reliable contraception methods are considered the following:

combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal or transdermal progestogen-only hormonal contraception associated with inhibition of ovulation oral, implanable or injectable intrauterine device (IUD) intrauterine hormone-releasing system (IUS) bilateral tubal occlusion vasectomised partner sexual abstinence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 36 hours post-administration
  Maximum plasma concentration, it is read directly from the raw data
AUC0-t | up to 36 hours post-administration
  Area under the plasma concentration curve from time 0 to the last measured

SECONDARY OUTCOMES:
AUC0-∞ | up to 36 hours post-administration
  Area under the plasma concentration-time curve extrapolated to infinity
Tmax | up to 36 hours post-administration
  Time until Cmax is reached, it is read directly from the observed concentrations
t1/2 | up to 36 hours post-administration
  Plasma concentration halflife, it is calculated from the ratio 0.693/λZ.
λz | up to 36 hours post-administration
  Terminal elimination rate constant, calculated from the slope of the final phase of the ln-concentration curve versus time with regression analysis
Residual area | up to 36 hours post-administration
  [AUC(0-∞)-AUC(0-t)]/AUC(0-∞)]

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Stefanidis, Professor, Principal Investigator — University of Thessaly Department of Medicine
Locations (1):
- BECRO Clinical Facility, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No